CLINICAL TRIAL: NCT00527709
Title: Hold Parameters on Likely Cardiovascular Depressant Medications (HOLD)
Brief Title: Hold Parameters on Likely Cardiovascular Depressant Medications
Status: Withdrawn | Type: Observational
Why Stopped: The study was a retrospective chart review and was mistakenly registered in ClinicalTrials.gov
Sponsor: Hackensack Meridian Health (Other)
Responsible Party: Sponsor
Other Study IDs: 06.01.025
Record Dates: First submitted 2007-09-07; First posted 2007-09-11 (Estimated); Last update posted 2020-08-05 (Actual); Status verified 2020-08

CONDITIONS: Asystole; Bradycardia; Hypotension
MeSH Terms: conditions — Heart Arrest; Bradycardia; Hypotension

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective

SUMMARY:
This pilot study is being pursued to observe whether certain medications are given to patients within a timeframe where their being given could play a part in a critical event in the management of the patient.

There are general rules about when it would be appropriate for these types of medications not to be given. However, it is not current standard practice for the criteria to be put in place without the expressed wishes of the ordering physician or their agent.

Research Question:

Can the administration of cardio-depressant medications be documented as a significant risk factor for hypotensive or bradycardic events?

ELIGIBILITY:
Inclusion Criteria:

* Serial evaluation of the first 50 documented events of Code Blue or call to Rapid Response Team involving hypotension, bradycardia or asystole in the adult inpatient population events beginning January 1, 2006.

Sex: All
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2006-08 (Actual); Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amit Tailor, MD, MBA, Principal Investigator — Hackensack Meridian Health
Locations (1):
- Hackensack University Medical Center, Hackensack, New Jersey, United States